CLINICAL TRIAL: NCT05492058
Title: Effects of Tactile Stimulus, Music Play and Virtual Reality Video Watching During Non-Stress Test on Maternal Anxiety and Fetal Parameters: A Randomized Controlled Clinical Trial
Brief Title: Tactile Stimulus, Music Play and Virtual Reality Video Watching During Non-Stress Test on Maternal Anxiety and Fetal Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Lokman Hekim University, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Lokman Hekim University
Record Dates: First submitted 2022-07-22; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Fetal Heart Failure; Fetal Movement Disorder
Keywords: nursing; fetal health; women; women health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- maternal touch (Experimental): maternal touch
  Interventions: Other: tactile stimulation group; Other: listen music; Other: virtual reality group
- music group (Experimental): music group
  Interventions: Other: tactile stimulation group; Other: listen music; Other: virtual reality group
- virtual reality group (Experimental): virtual reality group
  Interventions: Other: tactile stimulation group; Other: listen music; Other: virtual reality group
- control (No Intervention)

INTERVENTIONS:
Other: tactile stimulation group — The tactile stimulation group will be asked to touch their own abdomen during the NST procedure.
  Other Names: maternal touch
  Arms: maternal touch; music group; virtual reality group
Other: listen music — Pregnant women in the music group will listen to a song they want with headphones during the NST procedure.
  Other Names: music group
  Arms: maternal touch; music group; virtual reality group
Other: virtual reality group — Pregnant women in the virtual reality group will be shown a nature walk video with nature sounds (stream, bird, etc.) during the NST procedure.
  Arms: maternal touch; music group; virtual reality group

SUMMARY:
The research was carried out to determine the effects of tactile stimulation, music listening and virtual reality video watched during the non-stress test on maternal anxiety level and fetal parameters.

ELIGIBILITY:
Inclusion Criteria:

* - Not having any risk factors (pre-eclampsia, IUGG, premature rupture of membranes, getational diabetes, etc.) during pregnancy
* Absence of uterine contraction as a result of NST,
* No cardiovascular disease diagnosed in the fetus,
* Being in the 18-49 age group

Exclusion Criteria:

* Any complications in pregnancy and fetus
* Refusal to accept the final test

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Fetal heart rate, fetal movement | 20 minutes
  number
Maternal anxiety | 20 minutes
  STAI State Anxiety Inventory The emotions and behaviors expressed in the State Anxiety Inventory (STAI TX-I) items are answered by marking one of the options such as (1) never, (2) a little, (3) a lot, (4) completely, according to the severity of such experiences. The options in the Anxiety Scale are "almost never"(1), "sometimes"(2), "often"(3), "almost always"(4). Scoring ranges from 1 to 4. In the scale, there are direct or straight and reversed statements. Direct statements indicate negative emotions, reversed statements indicate positive emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman hekim University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No